CLINICAL TRIAL: NCT05242289
Title: Cytokine Adsorption in Lung Transplantation: a Randomized Controlled Pilot Study
Brief Title: Cytokine Adsorption in Lung Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University Hospital (Other)
Responsible Party: Principal Investigator, Sandra Lindstedt, Professor, Lund University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LUSorb
Record Dates: First submitted 2022-01-22; First posted 2022-02-16 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Lung Transplant Failure; Lung Transplant; Complications

STUDY DESIGN:
Intervention Model Description: The model consists of a randomized controlled pilot in human patients using a "cytokine adsorption" device.
  Lung transplant recipients are randomized to either the treatment group which undergoes cytokine adsorption using the medical device compared to the control group which has not received the cytokine adsorber.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treated (Active Comparator): Treatment using the medical "cytokine adsorption" device in conjunction with lung transplantation
  Interventions: Device: CytoSorb
- Non-treated (No Intervention): No additional treatment in conjunction with lung transplantation

INTERVENTIONS:
Device: CytoSorb — Medical device used hemoperfusion and cytokine adsorption in conjunction with lung transplantation.
  Arms: Treated

SUMMARY:
Lung transplantation (LTx) remains the gold standard for treating patients with irreversible end-stage pulmonary disease. Of the major organs transplanted, survival in LTx recipients remains the lowest (mean 5 years). Despite improvements, primary graft dysfunction (PGD), as defined by respiratory insufficiency and edema up to 72 hours post LTx, remains the leading cause of early mortality and contributes to the development of chronic lung allograft dysfunction (CLAD) which is the leading cause of late mortality (2). PGD develops within the first 72 hours after LTx. The development of CLAD increases quickly with cumulative incidence of 40-80 % within the first 3-5 years. There is a general lack of efficient treatments for PGD and CLAD. Prevention of PGD is therefore of crucial importance and has a direct impact on survival.

The present study is a randomized controlled pilot study which aims to compare patients undergoing LTx with and without the utilization of cytokine adsorption.

DETAILED DESCRIPTION:
Early intolerance to the newly transplanted lung starts at the time of transplantation and results in PGD driven by an intense inflammatory response. Cytokines play a critical role as signaling molecules that initiate, amplify, and maintain inflammatory responses both locally and systemically. The use of cytokine filtration devices to target middle- and low-molecular weight molecules has been shown to reduce levels of a diverse number of cytokines. These results have been demonstrated in the in vitro reduction of pathogen-associated molecular pattern molecules (PAMPS) and damage associated molecular patterns (DAMPS) as well as in in vivo studies involving orthotopic heart transplantation and kidney transplantation. Cytokine adsorption has been used successfully in clinical applications to both heart and kidney transplantation.

The present study is a randomized controlled pilot study which aims to collect preliminary data on the efficacy of a medical device through the comparison of patients undergoing LTx with and without cytokine adsorption.

ELIGIBILITY:
Inclusion Criteria:

* Double lung transplantation
* Single organ failure

Exclusion Criteria:

* Re-transplantation
* Drug abuse
* Kidney failure
* Liver failure
* Diabetes mellitus

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-03-02 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Oxygenation at 24 hours | 24 hours after lung transplantation
  Oxygenation expressed as the PaO2/FiO2 ratio at 24 hours
Oxygenation at 48 hours | 48 hours after lung transplantation
  Oxygenation expressed as the PaO2/FiO2 ratio at 48 hours
Oxygenation at 72 hours | 72 hours after lung transplantation
  Oxygenation expressed as the PaO2/FiO2 ratio at 72 hours

SECONDARY OUTCOMES:
Diffusion capacity of the lungs (DLCO) | 3 months after transplantation
  The primary function of the lungs is oxygenation of the blood and exhalation of carbon dioxide (CO2) from the blood. The ability of the lungs to perform this depends on a good alveolar ventilation, an even relationship between perfusion and ventilation, and good diffusion potential for oxygen (O2) and CO2 between alveolar, capillary and hemoglobin. This outcome will be measured through the diffusing capacity for carbon monoxide (DLCO)
Primary Graft dysfunction after 24 hours | 24 hours after lung transplantation
  Primary graft dysfunction (PGD) remains the leading cause of early mortality and contributes to the development of chronic lung allograft dysfunction (CLAD) which is the leading cause of late mortality. PGD develops over the first 72 hours after transplantation and is defined by evaluation of both the PaO2/FiO2 ratio and presence of lung edema on chest x-ray.
Primary Graft dysfunction after 48 hours | 48 hours after lungtransplantation
  PGD must also be assessed throughout the 72 hour period following completion of the transplantation and as such, this outcome will consist of the evaluation for PGD in the recipient 48 hours post-transplantation.
Primary Graft dysfunction after 72 hours | 72 hours after lungtransplantation
  PGD must also be assessed throughout the 72 hour period following completion of the transplantation and as such, this outcome will consist of the evaluation for PGD in the recipient 72 hours post-transplantation.
Urinary output as a measure of kidney function | First 3 months
  Kidney function is often impaired in transplant subjects due to the surgery itself but also secondary to drugs. The degree of acute kidney injury (AKI) can be assessed in part through measure of the urinary output.
Creatinine levels and clearance as a measure of kidney function | First 3 months
  To further assess the incidence of AKI, creatinine levels and its clearance will be measured.
Urea levels as a measure of kidney function | First 3 months
  Urea levels will also be measured to assess kidney function.
Rates of dialysis as a measure of kidney function | First 3 months
  The incidence of patients requiring dialysis will be also used to assess the frequency of AKI in the study population.
Volume blood loss | First 24 hours
  Given the nature of the transplantation itself as a major surgery, blood loss is expected after surgery and the volume of blood loss (mL) after surgery will be measured as a surgical outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Lindstedt, MD, PhD, Principal Investigator — Skånes universitetssjukhus Lund
Locations (1):
- Skåne University Hospital, Lund, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Niroomand A, Hirdman G, Olm F, Lindstedt S. Current Status and Future Perspectives on Machine Perfusion: A Treatment Platform to Restore and Regenerate Injured Lungs Using Cell and Cytokine Adsorption Therapy. Cells. 2021 Dec 29;11(1):91. doi: 10.3390/cells11010091. PMID 35011653
- [Result] Ghaidan H, Fakhro M, Lindstedt S. Impact of allograft ischemic time on long-term survival in lung transplantation: a Swedish monocentric study. Scand Cardiovasc J. 2020 Oct;54(5):322-329. doi: 10.1080/14017431.2020.1781240. Epub 2020 Jun 23. PMID 32573283
- [Result] Fakhro M, Ingemansson R, Skog I, Algotsson L, Hansson L, Koul B, Gustafsson R, Wierup P, Lindstedt S. 25-year follow-up after lung transplantation at Lund University Hospital in Sweden: superior results obtained for patients with cystic fibrosis. Interact Cardiovasc Thorac Surg. 2016 Jul;23(1):65-73. doi: 10.1093/icvts/ivw078. Epub 2016 Apr 6. PMID 27052747
- [Derived] Lindstedt S, Silverborn M, Lannemyr L, Pierre L, Larsson H, Grins E, Hyllen S, Dellgren G, Magnusson J. Design and Rationale of Cytokine Filtration in Lung Transplantation (GLUSorb): Protocol for a Multicenter Clinical Randomized Controlled Trial. JMIR Res Protoc. 2023 Dec 13;12:e52553. doi: 10.2196/52553. PMID 37855706
- See also: Pre print pre Clinical trail — https://www.researchsquare.com/article/rs-220294/v1